CLINICAL TRIAL: NCT02626169
Title: The Effect of Ticagrelor on 15-Epi-Lipoxin A4 and Inflammation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Pharmaceutical company sponsor withdrew support prior to enrollment of subjects.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Yochai Birnbaum, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-33860
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Atherosclerosis
Keywords: 15-epi-lipoxin A4; inflammation; atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): Clopidogrel 75 mg once a day by mouth for 30 days
  Interventions: Drug: Clopidogrel
- Ticagrelor (Active Comparator): Ticagrelor 90 mg twice daily by mouth for 30 days
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg once a day by mouth for 30 days
  Other Names: Plavix
  Arms: Clopidogrel
Drug: Ticagrelor — Ticagrelor 90 mg twice daily by mouth for 30 days
  Other Names: Brilinta
  Arms: Ticagrelor

SUMMARY:
Ticagrelor and clopidogrel are FDA-approved drugs for inhibition of platelet hyper-reactivity in certain clinical situations. The platelet inhibition and patient outcomes (PLATO) trial showed that in patients with acute coronary syndromes, ticagrelor significantly reduced the primary endpoint (cardiovascular death, myocardial infarction or stroke), all-cause mortality and cardiovascular mortality compared to clopidogrel. It has been suggested that in addition to its anti-platelet effects, ticagrelor has additional unique effects, including anti-inflammatory effects that are not shared by clopidogrel. In the present study the investigators will assess whether ticagrelor, as compared to clopidogrel, increases serum levels of 15-epi-lipoxin A4, a potent endogenous anti-inflammatory mediator.

DETAILED DESCRIPTION:
Clopidogrel, ticagrelor and prasugrel are routinely used for platelet inhibition in addition to aspirin in patients after acute coronary syndromes. The platelet inhibition and patient outcomes (PLATO) trial showed that in patients with acute coronary syndromes, ticagrelor significantly reduced the primary endpoint (cardiovascular death, myocardial infarction or stroke), all-cause mortality and cardiovascular mortality compared to clopidogrel. On the other hand, when compared with clopidogrel in patients with acute coronary syndromes with scheduled percutaneous coronary intervention, prasugrel therapy did not affect overall mortality despite the fact that it was associated with significantly reduced rates of ischemic events, including stent thrombosis, but with an increased risk of major bleeding, including fatal bleeding. This may suggest that ticagrelor possesses additional (pleiotropic) effects besides platelet inhibition.

The investigators have recently shown that pioglitazone increases 15-epi-lipoxin A4 blood levels in patients. The investigators have recently found that in the rat, ticagrelor increases tissue levels of 15-epi-lipoxin A4 in the heart, aorta and kidney.

It is plausible that some of the favorable effects of ticagrelor seen in the clinical studies are mediated via the anti-inflammatory effects of 15-epi-lipoxin A4.

15-epi-lipoxin A4 is a potent anti-inflammatory and inflammation-resolving mediator derived from arachidonic acid. Several studies have suggested that ticagrelor has anti-inflammatory properties in various animal models. In the present study the investigators will assess if ticagrelor increases blood 15-epi-lipoxin A4 levels at doses used in patients.

ELIGIBILITY:
Inclusion Criteria:

Provision of informed consent prior to any study specific procedures

Women of childbearing potential must be using an acceptable method of contraception to avoid pregnancy throughout the study

Patients with stable coronary artery disease (3-12 months after Acute Coronary Syndrome) who receive clopidogrel for at least 3 months.

Exclusion Criteria:

Recent stroke or acute coronary syndromes (<3 months before randomization).

Concurrent use of aspirin >100 mg/day where the dose reduction to 81 mg/day is contraindicated.

Current use of theophylline.

Concurrent use of Non Steroidal Anti-Inflammatory Drugs.

Patients receiving the following medications: ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, telithromycin, rifampin, dexamethasone, phenytoin, carbamazepine, or phenobarbital. Patients receiving simvastatin or lovastatin at doses greater than 40 mg daily.

Patients with type 2 diabetes with a fasting plasma glucose greater than 200 mg/dl.

Active inflammatory disease or chronic infection.

Contraindication for aspirin, clopidogrel or ticagrelor.

Women who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of 15-epi-lipoxin A4 | 30 days
  Percent change in plasma levels of 15-epi-lipoxin A4 from baseline (%)

SECONDARY OUTCOMES:
Plasma levels of C Reactive Protein (CRP) | 30 days
  Percent changes in plasma CRP from baseline (%)
platelet aggregation in blood sample | 30 days
  Percentage change in inhibition of platelet aggregation in blood sample from baseline (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Birnbaum, MD, Principal Investigator — Baylor College of Medicine, Houston
Locations (2):
- United States (2):
  - Baylor Clinic, Houston, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No